CLINICAL TRIAL: NCT00873093
Title: A Phase II Pilot Trial of Bortezomib (PS-341, Velcade) in Combination With Intensive Re-Induction Therapy for Children With Relapsed Acute Lymphoblastic Leukemia (ALL) and Lymphoblastic Lymphoma (LL)
Brief Title: Bortezomib and Combination Chemotherapy in Treating Young Patients With Relapsed Acute Lymphoblastic Leukemia or Lymphoblastic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01908; NCI-2011-01908 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AALL07P1 (Other: Children's Oncology Group); AALL07P1 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH)
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-11

CONDITIONS: B-cell Adult Acute Lymphoblastic Leukemia; B-cell Childhood Acute Lymphoblastic Leukemia; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Lymphoblastic Lymphoma; T-cell Adult Acute Lymphoblastic Leukemia; T-cell Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase; palmitoyl-L-asparaginase; Doxorubicin; Hydrocortisone; Vincristine; Cytarabine; Prednisone; Bortezomib; pegaspargase; Methotrexate; merphos; etoposide phosphate; Cyclophosphamide; Filgrastim; Granulocyte Colony-Stimulating Factor; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Pre-B ALL Relapse<18 mths from diagnosis (chemo) age<=21 yrs (Experimental): Re-Induction Block 1 patients receive vincristine sulfate, Prednisone, pegaspargase, Doxorubicin hydrochloride. Re-Induction Block 2 patients receive Cyclophosphamide, Etoposide phosphate, and Methotrexate. Re-Induction Block 3 patients receive Cytarabine.
  Interventions: Drug: L-asparaginase; Drug: doxorubicin hydrochloride; Drug: therapeutic hydrocortisone; Drug: vincristine sulfate; Drug: cytarabine; Drug: prednisone; Drug: bortezomib; Drug: pegaspargase; Drug: methotrexate; Drug: etoposide phosphate; Drug: cyclophosphamide; Biological: filgrastim; Drug: leucovorin calcium; Other: laboratory biomarker analysis; Drug: High Dose MTX
- Pre-B ALL Relapse 18-36 mths from diagnosis (chemo) age<=21 yr (Experimental): Re-Induction Block 1 patients receive vincristine sulfate, Prednisone, pegaspargase, Doxorubicin hydrochloride. Re-Induction Block 2 patients receive Cyclophosphamide, Etoposide phosphate, and Methotrexate. Re-Induction Block 3 patients receive Cytarabine.
  Interventions: Drug: L-asparaginase; Drug: doxorubicin hydrochloride; Drug: therapeutic hydrocortisone; Drug: vincristine sulfate; Drug: cytarabine; Drug: prednisone; Drug: bortezomib; Drug: pegaspargase; Drug: methotrexate; Drug: etoposide phosphate; Drug: cyclophosphamide; Biological: filgrastim; Drug: leucovorin calcium; Other: laboratory biomarker analysis; Drug: High Dose MTX
- Pre-B ALL Relapse<36 mths from diagnosis (chemo) age>21 yrs (Experimental): Re-Induction Block 1 patients receive vincristine sulfate, Prednisone, pegaspargase, Doxorubicin hydrochloride. Re-Induction Block 2 patients receive Cyclophosphamide, Etoposide phosphate, and Methotrexate. Re-Induction Block 3 patients receive Cytarabine.
  Interventions: Drug: L-asparaginase; Drug: doxorubicin hydrochloride; Drug: therapeutic hydrocortisone; Drug: vincristine sulfate; Drug: cytarabine; Drug: prednisone; Drug: bortezomib; Drug: pegaspargase; Drug: methotrexate; Drug: etoposide phosphate; Drug: cyclophosphamide; Biological: filgrastim; Drug: leucovorin calcium; Other: laboratory biomarker analysis; Drug: High Dose MTX
- T-cell ALL (Chemotherapy) (Experimental): Re-Induction Block 1 patients receive vincristine sulfate, Prednisone, pegaspargase, Doxorubicin hydrochloride. Re-Induction Block 2 patients receive Cyclophosphamide, Etoposide phosphate, and Methotrexate. Re-Induction Block 3 patients receive Cytarabine.
  Interventions: Drug: L-asparaginase; Drug: doxorubicin hydrochloride; Drug: therapeutic hydrocortisone; Drug: vincristine sulfate; Drug: cytarabine; Drug: prednisone; Drug: bortezomib; Drug: pegaspargase; Drug: methotrexate; Drug: etoposide phosphate; Drug: cyclophosphamide; Biological: filgrastim; Drug: leucovorin calcium; Other: laboratory biomarker analysis; Drug: High Dose MTX
- T-cell Lymphoblastic Lymphoma (LL) (Chemotherapy) (Experimental): Re-Induction Block 1 patients receive vincristine sulfate, Prednisone, pegaspargase, Doxorubicin hydrochloride. Re-Induction Block 2 patients receive Cyclophosphamide, Etoposide phosphate, and Methotrexate. Re-Induction Block 3 patients receive Cytarabine.
  Interventions: Drug: L-asparaginase; Drug: doxorubicin hydrochloride; Drug: therapeutic hydrocortisone; Drug: vincristine sulfate; Drug: cytarabine; Drug: prednisone; Drug: bortezomib; Drug: pegaspargase; Drug: methotrexate; Drug: etoposide phosphate; Drug: cyclophosphamide; Biological: filgrastim; Drug: leucovorin calcium; Other: laboratory biomarker analysis; Drug: High Dose MTX

INTERVENTIONS:
Drug: L-asparaginase — Given IM 6000 IU/m2/dose Days 2 and 9
  Other Names: ASNase; Colaspase; Crasnitin; Elspar; L-ASP
Drug: doxorubicin hydrochloride — Given IV 60 mg/m2/dose on Day 1
  Other Names: ADM; ADR; Adria
Drug: therapeutic hydrocortisone — Given IT (8mg - 15mg) Age-based dosing Block 1: Days 8,15, 22 and 29 Block 2: Days 1 and 22
  Other Names: Aeroseb-HC; Barseb HC; Cetacort; Cort-Dome; Cortef
Drug: vincristine sulfate — Given IV 1.5 mg/m2 (max 2 mg) on Days 1, 8, 15 and 22
  Other Names: liposomal vincristine; Marqibo; vincristine liposomal; vincristine sulfate liposome injection
Drug: cytarabine — Given IT or IV 3,000 mg/m2/dose on Days 1, 2, 8 and 9
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: prednisone — Given PO or IV 40 mg/m2/day on Days 1-28
  Other Names: DeCortin; Deltra
Drug: bortezomib — Given IV 1.3 mg/m2/dose Block 1: Days 1, 4, 8 and 11 Block 2: Days 1, 4 and 8
  Other Names: LDP 341; MLN341; VELCADE
Drug: pegaspargase — Given IM or IV (over 2 hours) 2500 IU/m2/dose on days 2, 8,15 and 22
  Other Names: L-asparaginase with polyethylene glycol; Oncaspar; PEG-ASP; PEG-L-asparaginase
Drug: methotrexate — Given IT (8mg - 15mg) Age-based dosing Block 1: Days 15 and 29 Block 2: Days 1 and 22
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Drug: etoposide phosphate — Given IV 100 mg/m2/dose on Days 1-5
  Other Names: ETOP; Etopophos
Drug: cyclophosphamide — Given IV 440 mg/m2/dose on Days 1-5
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Biological: filgrastim — Given IV or SC 5 micrograms/kg/dose Only on Day 6
  Other Names: G-CSF; Neupogen
Drug: leucovorin calcium — Given PO or IV 15mg/m2/dose q6h x 3 doses
  Other Names: CF; CFR; LV
Other: laboratory biomarker analysis — Correlative studies
Drug: High Dose MTX — IV 5000 mg/m2/dose Block 2: Day 22
  Other Names: methotrexate; amethopterin; Folex; methylaminopterin; Mexate

SUMMARY:
This pilot, phase II trial studies the side effects of giving bortezomib together with combination chemotherapy and to see how well it works in treating young patients with relapsed acute lymphoblastic leukemia or lymphoblastic lymphoma. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving bortezomib together with combination chemotherapy may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the toxicity, second complete response (CR2) rate at the end of Block 1 therapy, and 4-month event-free survival (EFS) for pediatric and young adult patients with relapsed acute lymphoblastic leukemia (ALL) treated with bortezomib in combination with intensive re-induction chemotherapy.

II. To evaluate bortezomib pharmacokinetics (PK) in patients receiving the combination regimen.

SECONDARY OBJECTIVES:

I. To assess minimal residual disease (MRD) in bone marrow following completion of each therapy block.

II. To assess the feasibility of measuring leukemia initiating cells (LIC) in patient samples before and after chemotherapy.

III. To discover biologic pathways associated with response and drug resistance using gene and protein expression profiles at baseline and following initial exposure to chemotherapy.

IV. To determine if bortezomib inhibits lymphoblast nuclear factor (NF)-kappa (k)-B activity in leukemia patients.

OUTLINE:

REINDUCTION BLOCK 1: Patients receive cytarabine intrathecally (IT) on day 1; vincristine sulfate IV over 1 minute on days 1, 8, 15, and 22; doxorubicin hydrochloride IV over 15 minutes on day 1; prednisone orally (PO) twice daily (BID) on days 1-28; bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11; and pegaspargase intramuscularly (IM) or IV over 1-2 hours on days 2, 8, 15, and 22. Patients with central nervous system (CNS)-negative disease (CNS1 or CNS2) also receive methotrexate IT on days 15 and 29; patients with CNS-positive disease (CNS3) receive triple intrathecal therapy (TIT) comprising methotrexate, hydrocortisone, and cytarabine IT on days 8, 15, 22, and 29. After completion of reinduction block 1, patients with ALL and M2 or M3 bone marrow proceed directly to reinduction block 2. Patients with ALL and M1 bone marrow or lymphoblastic lymphoma proceed to reinduction block 2 after blood counts recover. Patients with persistent cerebral spinal fluid (CSF) blasts after 6 doses of TIT or patients with progressive lymphoblastic lymphoma are removed from the study.

REINDUCTION BLOCK 2: Patients receive etoposide phosphate IV over 1-2 hours on days 1-5; cyclophosphamide IV over 15-30 minutes on days 1-5; bortezomib IV over 3-5 seconds on days 1, 4, and 8; filgrastim (G-CSF) subcutaneously (SC) or IV daily beginning on day 6 and continuing until blood counts recover*; high-dose methotrexate IV over 24 hours on day 22; and leucovorin calcium PO or IV every 6 hours on days 23 and 24. Patients with CNS-negative disease also receive methotrexate IT on days 1 and 22; patients with CNS-positive disease receive TIT on days 1 and 22. After completion of reinduction block 2, patients proceed to reinduction block 3 immediately or when blood counts recover. Patients with disease progression are removed from the study.

NOTE: *Patients do not receive G-CSF on day 8.

REINDUCTION BLOCK 3: Patients receive cytarabine IV over 3 hours BID on days 1, 2, 8, and 9; L-asparaginase IM on days 2 and 9; and G-CSF SC or IV daily beginning on day 10 and continuing until blood counts recover.

After completion of study treatment, patients are followed every 6 months for 3 years and then annually for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis

  * Pre-B ALL in first early (< 36 months from diagnosis) isolated bone marrow (BM) or combined BM/extramedullary relapse; or
  * T-cell ALL in first isolated BM or combined relapse; or
  * T-LL in first relapse
* Patients with leukemia must have had histologic verification of the malignancy at relapse, including immunophenotyping to confirm diagnosis
* Patients with lymphoblastic lymphoma must have measurable disease documented by clinical, radiographic, or histologic criteria; patients must have relapsed or become refractory to conventional therapy
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2; use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* Patients who relapse while receiving standard ALL maintenance chemotherapy will not be required to have a waiting period before entry onto this study
* Patients who relapse on therapy other than standard ALL maintenance therapy must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study
* At least 14 days since the completion of cytotoxic therapy with the exception of hydroxyurea, which is permitted up to 24 hours prior to the start of protocol therapy
* At least 7 days since the completion of therapy with a biologic agent or donor lymphocyte infusions (DLI); for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur
* No evidence of active graft-vs-host disease (GVHD) and >= 4 months must have elapsed; must not be receiving GVHD prophylaxis
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * 1 month to < 6 months (0.4 male, 0.4 female)
  * 6 months to < 1 year (0.5 male, 0.5 female)
  * 1 to < 2 years (0.6 male, 0.6 female)
  * 2 to < 6 years (0.8 male, 0.8 female)
  * 6 to < 10 years (1 male, 1 female)
  * 10 to < 13 years (1.2 male, 1.2 female)
  * 13 to < 16 years (1.5 male, 1.4 female)
  * >= 16 years (1.7 male, 1.4 female)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 3 x ULN for age, unless elevation due to leukemia infiltration
* Shortening fraction of >= 27% by echocardiogram, or
* Ejection fraction of >= 50% by gated radionuclide study
* No evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry >= 94% at sea level (> 90% if at high altitude)
* No evidence of acute pulmonary infiltrates on chest radiograph
* Patients with seizure disorder may be enrolled if on allowed anticonvulsants and well controlled; benzodiazepines and gabapentin are acceptable
* Central nervous system (CNS) toxicity =< grade 2
* Peripheral nervous system (PNS) toxicity < grade 3
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, FDA, and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients with Philadelphia chromosome positive ALL are not eligible unless refractory to at least one tyrosine kinase inhibitor (TKI) therapy; patients that are unable to tolerate TKI therapy due to toxicity are eligible
* Patients with mature B-cell ALL, ie, leukemia with B-cell (soluble immunoglobulin [sIg] positive and kappa or lambda restricted positivity) ALL, with French-American-British (FAB) L3 morphology and/or a myc translocation, are not eligible
* Extramedullary disease status: patients with isolated CNS disease or isolated testicular disease are not eligible
* Patients with known optic nerve and/or retinal involvement are not eligible; patients presenting with visual disturbances should have an ophthalmological exam and, if indicated, an magnetic resonance imaging (MRI) to determine optic nerve or retinal involvement
* Patients with concomitant genetic syndrome: patients with Down syndrome, Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome are not eligible
* Cumulative prior anthracycline exposure must not exceed 400 mg/m^2
* Patients taking anticonvulsants known to activate the cytochrome p450 system, in particular anticonvulsants such as phenytoin, carbamazepine, and phenobarbital, are not eligible; benzodiazepines and gabapentin are acceptable
* Patients who have previously received bortezomib or other proteasome inhibitors are not eligible
* Patients who have a known allergy to doxorubicin, cytarabine, both etoposide and etopophos, boron, mannitol or bortezomib are not eligible
* Patients who cannot receive any asparaginase products (E. Coli, PEG-asparaginase, or Erwinia asparaginase) on this study (eg, due to prior severe pancreatitis, stroke or other toxicity) are not eligible; patients who initially receive asparaginase, but must discontinue due to toxicity, remain eligible; patients with clinically significant prior allergies to pegaspargase are eligible if Erwinia L-asparaginase can be substituted
* Patients who are pregnant or breast-feeding are not eligible for this study; negative pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective birth control method
* Patients must not have received any prior re-induction attempts and must not have received treatment for prior extramedullary relapse; patients with primary induction failure are not eligible

Ages: 1 Year to 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 148 (Actual)
Dates: Start 2009-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terzah Horton, MD PhD, Principal Investigator — Children's Oncology Group
Locations (171):
- United States (157):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - City of Hope Medical Center, Duarte, California
  - City of Hope, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Childrens Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California at Davis Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - University of California San Francisco Medical Center-Parnassus, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lombardi Comprehensive Cancer Center at Georgetown University, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Memorial Healthcare System - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville South, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph Children's Hospital of Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Services, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Floating Hospital for Children at Tufts Medical Center, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Columbia Regional, Columbia, Missouri
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - UMDNJ - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of New Mexico, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - New York University Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health Richland, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Science Center-Amarillo, Amarillo, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Childrens Hospital-King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Carilion Clinic Children's Hospital, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston, Charleston, West Virginia
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (12):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Chedoke-McMaster Hospitals, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- San Jorge Children's Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Horton TM, Whitlock JA, Lu X, O'Brien MM, Borowitz MJ, Devidas M, Raetz EA, Brown PA, Carroll WL, Hunger SP. Bortezomib reinduction chemotherapy in high-risk ALL in first relapse: a report from the Children's Oncology Group. Br J Haematol. 2019 Jul;186(2):274-285. doi: 10.1111/bjh.15919. Epub 2019 Apr 7. PMID 30957229
- [Derived] Hanley MJ, Mould DR, Taylor TJ, Gupta N, Suryanarayan K, Neuwirth R, Esseltine DL, Horton TM, Aplenc R, Alonzo TA, Lu X, Milton A, Venkatakrishnan K. Population Pharmacokinetic Analysis of Bortezomib in Pediatric Leukemia Patients: Model-Based Support for Body Surface Area-Based Dosing Over the 2- to 16-Year Age Range. J Clin Pharmacol. 2017 Sep;57(9):1183-1193. doi: 10.1002/jcph.906. Epub 2017 Apr 18. PMID 28419486

RESULTS

PARTICIPANT FLOW:
Groups:
- Pre-B ALL Relapse<36 Mths From Diagnosis (Chemo) Age>21 yr; Pre-B ALL Relapse 18-36 Mths From Diagnosis (Chemo) Age<=21 yr; Pre-B ALL Relapse<18 Mths From Diagnosis (Chemo) Age<=21 Yrs; T-cell ALL (Chemotherapy); T-cell Lymphoblastic Lymphoma (LL) (Chemotherapy): Re-Induction Block 1 patients receive liposomal vincristine sulfate , Prednisone, pegaspargase and Doxorubicin hydrochloride. Re-Induction Block 2 patients receive Cyclophosphamide, Etoposide phosphate, and Methotrexate. Re-Induction Block 3 patients receive Cytarabine and L-Asparaginase. Patients receive Bortezomib on days 1, 4, 8 & 11 of Block 1 and days 1, 4, & 8 of Block 2.
Period: Overall Study
Arm/Group | Pre-B ALL Relapse<36 Mths From Diagnosis (Chemo) Age>21 yr | Pre-B ALL Relapse 18-36 Mths From Diagnosis (Chemo) Age<=21 yr | Pre-B ALL Relapse<18 Mths From Diagnosis (Chemo) Age<=21 Yrs | T-cell ALL (Chemotherapy) | T-cell Lymphoblastic Lymphoma (LL) (Chemotherapy)
Started | 4 | 62 | 49 | 23 | 10
Completed | 3 | 35 | 33 | 12 | 8
Not Completed | 1 | 27 | 16 | 11 | 2
Not completed — Adverse Event | 0 | 2 | 0 | 0 | 0
Not completed — Death | 0 | 3 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 17 | 10 | 10 | 2
Not completed — Withdrawal by Subject | 1 | 4 | 4 | 0 | 0
Not completed — Ineligible | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pre-B ALL Relapse < 36 Mths From Dx (Chemotherapy) Age >21 Yrs; Pre-B ALL Relapse 18-36 Mths From Dx (Chemotherapy)Age<=21 Yrs; Pre-B ALL Relapse <18 Mths From Dx (Chemotherapy) Age <=21 Yrs; T-cell ALL (Chemotherapy); T-cell Lymphoblastic Lymphoma (LL) (Chemotherapy): Re-Induction Block 1 patients receive liposomal vincristine sulfate , Prednisone, pegaspargase and Doxorubicin hydrochloride. Re-Induction Block 2 patients receive Cyclophosphamide, Etoposide phosphate, and Methotrexate. Re-Induction Block 3 patients receive Cytarabine and L-Asparaginase. Patients receive Bortezomib on days 1, 4, 8 & 11 of Block 1 and days 1, 4, & 8 of Block 2.
- Total: Total of all reporting groups
Arm/Group | Pre-B ALL Relapse < 36 Mths From Dx (Chemotherapy) Age >21 Yrs | Pre-B ALL Relapse 18-36 Mths From Dx (Chemotherapy)Age<=21 Yrs | Pre-B ALL Relapse <18 Mths From Dx (Chemotherapy) Age <=21 Yrs | T-cell ALL (Chemotherapy) | T-cell Lymphoblastic Lymphoma (LL) (Chemotherapy) | Total
Number analyzed (Participants) | 4 | 62 | 49 | 23 | 10 | 148
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 53 | 45 | 20 | 8 | 126
  Between 18 and 65 years | 4 | 9 | 4 | 3 | 2 | 22
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.14 (0.57) | 10.16 (5.77) | 9.27 (6.06) | 13.00 (5.28) | 13.79 (6.27) | 10.91 (6.23)
Gender [Count of Participants; unit: Participants]
  Female | 2 | 29 | 21 | 6 | 5 | 63
  Male | 2 | 33 | 28 | 17 | 5 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 15 | 18 | 4 | 0 | 38
  Not Hispanic or Latino | 3 | 44 | 31 | 19 | 10 | 107
  Unknown or Not Reported | 0 | 3 | 0 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 1 | 0 | 3
  Asian | 0 | 3 | 1 | 1 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1 | 2
  Black or African American | 0 | 9 | 8 | 4 | 1 | 22
  White | 2 | 44 | 34 | 16 | 8 | 104
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 5 | 5 | 1 | 0 | 12

OUTCOME MEASURES:

1. Primary Outcome: Second Complete Remission Rate at the End of Block 1 Reinduction Chemotherapy
Description: The percentage of eligible and evaluable patients who have achieved complete response at the end Block 1 of re-induction therapy.
Time Frame: The outcome is measured the end of Block 1 (Day 36 of Block 1) of re-induction therapy.
Population: The analysis on this primary outcome is limited to pre-B ALL with age <= 21 years who relapsed < 36 months only (stratum 1 & 2) per protocol section 9.2.1.
Measure: Number; unit: Percentage of participants
Arm/Group | Pre-B ALL Relapse < 36 Mths From Dx (Chemotherapy) Age >21 Yrs | Pre-B ALL Relapse 18-36 Mths From Dx (Chemotherapy)Age<=21 Yrs | Pre-B ALL Relapse <18 Mths From Dx (Chemotherapy) Age <=21 Yrs | T-cell ALL (Chemotherapy) | T-cell Lymphoblastic Lymphoma (LL) (Chemotherapy)
Number analyzed (Participants) | 0 | 54 | 46 | 0 | 0
Percentage of participants |  | 72.2 | 63 |  |

2. Primary Outcome: Event Free Survival
Description: Percentage of patients who were event free at 4 months
Time Frame: 4 months after enrollment
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Pre-B ALL Relapse < 36 Mths From Dx (Chemotherapy) Age >21 Yrs | Pre-B ALL Relapse 18-36 Mths From Dx (Chemotherapy)Age<=21 Yrs | Pre-B ALL Relapse <18 Mths From Dx (Chemotherapy) Age <=21 Yrs | T-cell ALL (Chemotherapy) | T-cell Lymphoblastic Lymphoma (LL) (Chemotherapy)
Number analyzed (Participants) | 0 | 54 | 46 | 0 | 0
Percentage of participants |  | 68.5 | 37.8 |  |

3. Primary Outcome: Toxic Death Rate
Description: The proportion of toxic death rate among all eligible patients.
Time Frame: 4 months
Population: The toxic death was monitored for all eligible patients. It was not compared between subgroups per protocol 9.3.2.
Measure: Number; unit: percentage of participants
Groups:
- Overall: All enrolled eligible patients.
Arm/Group | Overall
Number analyzed (Participants) | 146
percentage of participants | 2.1

4. Primary Outcome: Severe Adverse Events (SAE) Rate.
Description: The proportion of SAE rate among all eligible patients
Time Frame: 4 months
Population: The SAE event was monitored for all eligible patients. It was not compared between subgroups per protocol 9.3.2.
Measure: Number; unit: percentage of participants
Arm/Group | Overall
Number analyzed (Participants) | 146
percentage of participants | 8.2

5. Secondary Outcome: Rate of Minimal Residual Disease (MRD) < 0.01% at End Block 1
Description: Percentage of eligible and evaluable patients with MRD < 0.01% among those who had successful MRD determination at the end of Block 1.
Time Frame: End of Block 1 (Day 36 of Block 1) of re-induction therapy
Population: The MRD analysis is limited to eligible and evaluable pre-B ALL with age <= 21 years who relapsed < 36 months only (stratum 1 & 2) and have successful MRD determination at the end of Block 1per protocol section 9.3.3.
Measure: Number; unit: percentage of participants
Arm/Group | Pre-B ALL Relapse < 36 Mths From Dx (Chemotherapy) Age >21 Yrs | Pre-B ALL Relapse 18-36 Mths From Dx (Chemotherapy)Age<=21 Yrs | Pre-B ALL Relapse <18 Mths From Dx (Chemotherapy) Age <=21 Yrs | T-cell ALL (Chemotherapy) | T-cell Lymphoblastic Lymphoma (LL) (Chemotherapy)
Number analyzed (Participants) | 0 | 48 | 40 | 0 | 0
percentage of participants |  | 35.4 | 25 |  |

6. Secondary Outcome: Rate of Minimal Residual Disease (MRD) < 0.01% at End Block 2
Description: Percentage of eligible and evaluable patients with MRD < 0.01% among those who had successful MRD determination at the end of Block 2.
Time Frame: End of Block 2 (Day 36 of Block 2) of re-induction therapy
Population: The MRD analysis is limited to eligible and evaluable pre-B ALL with age <= 21 years who relapsed < 36 months only (stratum 1 & 2) and have successful MRD determination at the end of Block 2per protocol section 9.3.3.
Measure: Number; unit: percentage of participants
Arm/Group | Pre-B ALL Relapse < 36 Mths From Dx (Chemotherapy) Age >21 Yrs | Pre-B ALL Relapse 18-36 Mths From Dx (Chemotherapy)Age<=21 Yrs | Pre-B ALL Relapse <18 Mths From Dx (Chemotherapy) Age <=21 Yrs | T-cell ALL (Chemotherapy) | T-cell Lymphoblastic Lymphoma (LL) (Chemotherapy)
Number analyzed (Participants) | 0 | 30 | 19 | 0 | 0
percentage of participants |  | 66.7 | 42.1 |  |

7. Secondary Outcome: Rate of Minimal Residual Disease (MRD) < 0.01% at End Block 3
Description: Percentage of eligible and evaluable patients with MRD < 0.01% among those who had successful MRD determination at the end of Block 3.
Time Frame: End of Block 3 (Day 36 of Block 3) of re-induction therapy
Population: The MRD analysis is limited to eligible and evaluable pre-B ALL with age <= 21 years who relapsed < 36 months only (stratum 1 & 2) and have successful MRD determination at the end of Block 3per protocol section 9.3.3.
Measure: Number; unit: Percentage of participants
Arm/Group | Pre-B ALL Relapse < 36 Mths From Dx (Chemotherapy) Age >21 Yrs | Pre-B ALL Relapse 18-36 Mths From Dx (Chemotherapy)Age<=21 Yrs | Pre-B ALL Relapse <18 Mths From Dx (Chemotherapy) Age <=21 Yrs | T-cell ALL (Chemotherapy) | T-cell Lymphoblastic Lymphoma (LL) (Chemotherapy)
Number analyzed (Participants) | 0 | 20 | 11 | 0 | 0
Percentage of participants |  | 80 | 63.6 |  |

8. Other Pre Specified Outcome: NF-kB Activity
Description: NF-kB activity will be measured as a continuous variable (ng NF-kB/ug protein). Differences in NF-kB activity between time points will be assessed using summary statistics such as mean, standard deviation, and range.
Time Frame: Up to 5 years
Population: These were for correlative biology studies and the data were not collected in COG database.
Groups:
- Pre-B ALL Relapse < 36 Mths From Dx (Chemotherapy) Age >21 Yrs: Re-Induction Block 1 patients receive vincristine sulfate, Prednisone, pegaspargase, Doxorubicin hydrochloride. Re-Induction Block 2 patients receive Cyclophosphamide, Etoposide phosphate, and MTX. Re-Induction Block 3 patients receive Cytarabine.
  L-asparaginase: Given IM 6000 IU/m2/dose Days 2 and 9
  doxorubicin hydrochloride: Given IV 60 mg/m2/dose on Day 1
  therapeutic hydrocortisone: Given IT (8mg - 15mg) Age-based dosing Block 1: Days 8,15, 22 & 29 Block 2: Days 1 & 22
  vincristine sulfate: Given IV 1.5 mg/m2 (max 2 mg) on Days 1, 8, 15 and 22
  cytarabine: Given IT or IV 3,000 mg/m2/dose on Days 1, 2, 8 & 9
  prednisone: Given PO or IV 40 mg/m2/day on Days 1-28
  bortezomib: Given IV 1.3 mg/m2/dose Block 1: Days 1, 4, 8 & 11 Block 2: Days 1, 4 & 8
  pegaspargase: Given IM or IV (over 2 hours) 2500 IU/m2/dose on days 2, 8,15 & 22
  MTX: Given IT (8mg - 15mg) Age-based dosing Block 1: Days 15 & 29 Block 2: Days 1 & 22
  etopo
- Pre-B ALL Relapse 18-36 Mths From Dx (Chemotherapy)Age<=21 Yrs; T-cell Lymphoblastic Lymphoma (LL) (Chemotherapy): Re-Induction Block 1 patients receive vincristine sulfate, Prednisone, pegaspargase, Doxorubicin hydrochloride. Re-Induction Block 2 patients receive Cyclophosphamide, Etoposide phosphate, and MTX. Re-Induction Block 3 patients receive Cytarabine.
  L-asparaginase: Given IM 6000 IU/m2/dose Days 2 & 9
  doxorubicin hydrochloride: Given IV 60 mg/m2/dose on Day 1
  therapeutic hydrocortisone: Given IT (8mg - 15mg) Age-based dosing Block 1: Days 8,15, 22 & 29 Block 2: Days 1 & 22
  vincristine sulfate: Given IV 1.5 mg/m2 (max 2 mg) on Days 1, 8, 15 & 22
  cytarabine: Given IT or IV 3,000 mg/m2/dose on Days 1, 2, 8 & 9
  prednisone: Given PO or IV 40 mg/m2/day on Days 1-28
  bortezomib: Given IV 1.3 mg/m2/dose Block 1: Days 1, 4, 8 & 11 Block 2: Days 1, 4 & 8
  pegaspargase: Given IM or IV (over 2 hours) 2500 IU/m2/dose on days 2, 8,15 & 22
  MTX: Given IT (8mg - 15mg) Age-based dosing Block 1: Days 15 & 29 Block 2: Days 1 & 22
  etopo
- Pre-B ALL Relapse <18 Mths From Dx (Chemotherapy) Age <=21 Yrs: Re-Induction Block 1 patients receive vincristine sulfate, Prednisone, pegaspargase, Doxorubicin hydrochloride. Re-Induction Block 2 patients receive Cyclophosphamide, Etoposide phosphate, and Methotrexate. Re-Induction Block 3 patients receive Cytarabine.
  L-asparaginase: Given IM 6000 IU/m2/dose Days 2 & 9
  doxorubicin hydrochloride: Given IV 60 mg/m2/dose on Day 1
  therapeutic hydrocortisone: Given IT (8mg - 15mg) Age-based dosing Block 1: Days 8,15, 22 & 29 Block 2: Days 1 & 22
  vincristine sulfate: Given IV 1.5 mg/m2 (max 2 mg) on Days 1, 8, 15 & 22
  cytarabine: Given IT or IV 3,000 mg/m2/dose on Days 1, 2, 8 & 9
  prednisone: Given PO or IV 40 mg/m2/day on Days 1-28
  bortezomib: Given IV 1.3 mg/m2/dose Block 1: Days 1, 4, 8 & 11 Block 2: Days 1, 4 & 8
  pegaspargase: Given IM or IV (over 2 hours) 2500 IU/m2/dose on days 2, 8,15 & 22
  MTX: Given IT (8mg - 15mg) Age-based dosing Block 1: Days 15 & 29 Block 2: Days 1 & 22
  etopo
- T-cell ALL (Chemotherapy): Re-Induction Block 1 patients receive vincristine sulfate, Prednisone, pegaspargase, Doxorubicin hydrochloride. Re-Induction Block 2 patients receive Cyclophosphamide, Etoposide phosphate, and Methotrexate. Re-Induction Block 3 patients receive Cytarabine.
  L-asparaginase: Given IM 6000 IU/m2/dose Days 2 & 9
  doxorubicin hydrochloride: Given IV 60 mg/m2/dose on Day 1
  therapeutic hydrocortisone: Given IT (8mg - 15mg) Age-based dosing Block 1: Days 8,15, 22 & 29 Block 2: Days 1 & 22
  vincristine sulfate: Given IV 1.5 mg/m2 (max 2 mg) on Days 1, 8, 15 & 22
  cytarabine: Given IT or IV 3,000 mg/m2/dose on Days 1, 2, 8 & 9
  prednisone: Given PO or IV 40 mg/m2/day on Days 1-28
  bortezomib: Given IV 1.3 mg/m2/dose Block 1: Days 1, 4, 8 & 11 Block 2: Days 1, 4 & 8
  pegaspargase: Given IM or IV (over 2 hours) 2500 IU/m2/dose on days 2, 8,15 & 22
  methotrexate: Given IT (8mg - 15mg) Age-based dosing Block 1: Days 15 & 29 Block 2: Days 1 & 22
  etopo
Arm/Group | Pre-B ALL Relapse < 36 Mths From Dx (Chemotherapy) Age >21 Yrs | Pre-B ALL Relapse 18-36 Mths From Dx (Chemotherapy)Age<=21 Yrs | Pre-B ALL Relapse <18 Mths From Dx (Chemotherapy) Age <=21 Yrs | T-cell ALL (Chemotherapy) | T-cell Lymphoblastic Lymphoma (LL) (Chemotherapy)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

9. Other Pre Specified Outcome: Expression of Apoptotic and Cell Cycle Proteins Assessed by Using Gene and Tissue Microarrays and Immunoblots
Description: Characterized using descriptive statistics. If differences are noted between pre- and post-treatment protein expression, pairwise comparisons will be made using paired t-test or an equivalent nonparametric test. The normality assumption will be assessed on the log-transformed data prior to paired t-test evaluation.
Time Frame: Up to 5 years
Population: These were for correlative biology studies and the data were not collected in COG database.
Groups:
- Pre-B ALL Relapse < 36 Mths From Dx (Chemotherapy) Age >21 Yrs: Re-Induction Block 1 patients receive vincristine sulfate, Prednisone, pegaspargase, Doxorubicin hydrochloride. Re-Induction Block 2 patients receive Cyclophosphamide, Etoposide phosphate and MTX. Re-Induction Block 3 patients receive Cytarabine.
  L-asparaginase: Given IM 6000 IU/m2/dose Days 2 and 9
  doxorubicin hydrochloride: Given IV 60 mg/m2/dose on Day 1
  therapeutic hydrocortisone: Given IT (8mg - 15mg) Age-based dosing Block 1: Days 8,15, 22 & 29 Block 2: Days 1 & 22
  vincristine sulfate: Given IV 1.5 mg/m2 (max 2 mg) on Days 1, 8, 15 and 22
  cytarabine: Given IT or IV 3,000 mg/m2/dose on Days 1, 2, 8 & 9
  prednisone: Given PO or IV 40 mg/m2/day on Days 1-28
  bortezomib: Given IV 1.3 mg/m2/dose Block 1: Days 1, 4, 8 & 11 Block 2: Days 1, 4 & 8
  pegaspargase: Given IM or IV (over 2 hours) 2500 IU/m2/dose on days 2, 8,15 & 22
  MTX: Given IT (8mg - 15mg) Age-based dosing Block 1: Days 15 & 29 Block 2: Days 1 & 22
  etopo
- Pre-B ALL Relapse 18-36 Mths From Dx (Chemotherapy)Age<=21 Yrs: Re-Induction Block 1 patients receive vincristine sulfate, Prednisone, pegaspargase, Doxorubicin hydrochloride. Re-Induction Block 2 patients receive Cyclophosphamide, Etoposide phosphate and MTX. Re-Induction Block 3 patients receive Cytarabine.
  L-asparaginase: Given IM 6000 IU/m2/dose Days 2 & 9
  doxorubicin hydrochloride: Given IV 60 mg/m2/dose on Day 1
  therapeutic hydrocortisone: Given IT (8mg - 15mg) Age-based dosing Block 1: Days 8,15, 22 & 29 Block 2: Days 1 & 22
  vincristine sulfate: Given IV 1.5 mg/m2 (max 2 mg) on Days 1, 8, 15 & 22
  cytarabine: Given IT or IV 3,000 mg/m2/dose on Days 1, 2, 8 & 9
  prednisone: Given PO or IV 40 mg/m2/day on Days 1-28
  bortezomib: Given IV 1.3 mg/m2/dose Block 1: Days 1, 4, 8 & 11 Block 2: Days 1, 4 & 8
  pegaspargase: Given IM or IV (over 2 hours) 2500 IU/m2/dose on days 2, 8,15 & 22
  MTX: Given IT (8mg - 15mg) Age-based dosing Block 1: Days 15 & 29 Block 2: Days 1 & 22
  etopo
- Pre-B ALL Relapse <18 Mths From Dx (Chemotherapy) Age <=21 Yrs; T-cell Lymphoblastic Lymphoma (LL) (Chemotherapy): Re-Induction Block 1 patients receive vincristine sulfate, Prednisone, pegaspargase, Doxorubicin hydrochloride. Re-Induction Block 2 patients receive Cyclophosphamide, Etoposide phosphate, and MTX. Re-Induction Block 3 patients receive Cytarabine.
  L-asparaginase: Given IM 6000 IU/m2/dose Days 2 & 9
  doxorubicin hydrochloride: Given IV 60 mg/m2/dose on Day 1
  therapeutic hydrocortisone: Given IT (8mg - 15mg) Age-based dosing Block 1: Days 8,15, 22 & 29 Block 2: Days 1 & 22
  vincristine sulfate: Given IV 1.5 mg/m2 (max 2 mg) on Days 1, 8, 15 & 22
  cytarabine: Given IT or IV 3,000 mg/m2/dose on Days 1, 2, 8 & 9
  prednisone: Given PO or IV 40 mg/m2/day on Days 1-28
  bortezomib: Given IV 1.3 mg/m2/dose Block 1: Days 1, 4, 8 & 11 Block 2: Days 1, 4 & 8
  pegaspargase: Given IM or IV (over 2 hours) 2500 IU/m2/dose on days 2, 8,15 & 22
  MTX: Given IT (8mg - 15mg) Age-based dosing Block 1: Days 15 & 29 Block 2: Days 1 & 22
  etopo
- T-cell ALL (Chemotherapy): Re-Induction Block 1 patients receive vincristine sulfate, Prednisone, pegaspargase, Doxorubicin hydrochloride. Re-Induction Block 2 patients receive Cyclophosphamide, Etoposide phosphate, and MTX. Re-Induction Block 3 patients receive Cytarabine.
  L-asparaginase: Given IM 6000 IU/m2/dose Days 2 & 9
  doxorubicin hydrochloride: Given IV 60 mg/m2/dose on Day 1
  therapeutic hydrocortisone: Given IT (8mg - 15mg) Age-based dosing Block 1: Days 8,15, 22 & 29 Block 2: Days 1 & 22
  vincristine sulfate: Given IV 1.5 mg/m2 (max 2 mg) on Days 1, 8, 15 & 22
  cytarabine: Given IT or IV 3,000 mg/m2/dose on Days 1, 2, 8 & 9
  prednisone: Given PO or IV 40 mg/m2/day on Days 1-28
  bortezomib: Given IV 1.3 mg/m2/dose Block 1: Days 1, 4, 8 & 11 Block 2: Days 1, 4 & 8
  pegaspargase: Given IM or IV (over 2 hours) 2500 IU/m2/dose on days 2, 8,15 & 22
  methotrexate: Given IT (8mg - 15mg) Age-based dosing Block 1: Days 15 & 29 Block 2: Days 1 & 22
  etopo
Arm/Group | Pre-B ALL Relapse < 36 Mths From Dx (Chemotherapy) Age >21 Yrs | Pre-B ALL Relapse 18-36 Mths From Dx (Chemotherapy)Age<=21 Yrs | Pre-B ALL Relapse <18 Mths From Dx (Chemotherapy) Age <=21 Yrs | T-cell ALL (Chemotherapy) | T-cell Lymphoblastic Lymphoma (LL) (Chemotherapy)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

10. Other Pre Specified Outcome: Change in Stem Cell Percentage
Description: Will use descriptive statistics to assess mean +/- standard deviation for stem cell percentage before and after bortezomib treatment. If there appears to be a difference in responders vs. non-responders, stem cell percentage differences between responders and non-responders will be compared using a paired t-test or equivalent nonparametric test.
Time Frame: Baseline to post-treatment with bortezomib
Population: These were for correlative biology studies and the data were not collected in COG database.
Arm/Group | Pre-B ALL Relapse < 36 Mths From Dx (Chemotherapy) Age >21 Yrs | Pre-B ALL Relapse 18-36 Mths From Dx (Chemotherapy)Age<=21 Yrs | Pre-B ALL Relapse <18 Mths From Dx (Chemotherapy) Age <=21 Yrs | T-cell ALL (Chemotherapy) | T-cell Lymphoblastic Lymphoma (LL) (Chemotherapy)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

11. Other Pre Specified Outcome: Plasma Concentration-time Profiles
Description: Will be analyzed using descriptive statistics and will be graphically displayed by age group and stratum. PK data will be analyzed using methods such as nonlinear mixed effects modeling to estimate bortezomib clearance and volume of distribution (and the associated 95% confidence intervals) in each age group (2-11 years and 12-16 years of age).
Time Frame: Up to day 8 of block 2
Population: These were for correlative biology studies and the data were not collected in COG database.
Arm/Group | Pre-B ALL Relapse < 36 Mths From Dx (Chemotherapy) Age >21 Yrs | Pre-B ALL Relapse 18-36 Mths From Dx (Chemotherapy)Age<=21 Yrs | Pre-B ALL Relapse <18 Mths From Dx (Chemotherapy) Age <=21 Yrs | T-cell ALL (Chemotherapy) | T-cell Lymphoblastic Lymphoma (LL) (Chemotherapy)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

12. Other Pre Specified Outcome: Pharmacokinetics (PK) of Bortezomib in Patients Receiving Multi-agent Combination Therapy.
Description: This outcome measure cannot be reported due to the data used for analysis was not collected.
Time Frame: Day 8 of blocks 1 and 2
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: SAE field contains NCI CTCAEs submitted via expedited reporting (NCI AdEERs/CAeRs). AE field contains grade 3 & higher CTCAEs reported on study excluding reported SAEs. Analyses on outcomes was based on eligible & evaluable patients. Reported AEs should be enrolled eligible patient based, so numbers of participants in the two AE tables are larger.
Arm/Group | Pre-B ALL Relapse < 36 Mths From Dx (Chemotherapy) Age >21 Yrs | Pre-B ALL Relapse 18-36 Mths From Dx (Chemotherapy)Age<=21 Yrs | Pre-B ALL Relapse <18 Mths From Dx (Chemotherapy) Age <=21 Yrs | T-cell ALL (Chemotherapy) | T-cell Lymphoblastic Lymphoma (LL) (Chemotherapy)
Serious Adverse Events (participants affected / at risk) | 2/4 | 47/61 | 40/49 | 18/22 | 7/10
Other Adverse Events (participants affected / at risk) | 4/4 | 58/61 | 44/49 | 21/22 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-B ALL Relapse < 36 Mths From Dx (Chemotherapy) Age >21 Yrs (N=4) | Pre-B ALL Relapse 18-36 Mths From Dx (Chemotherapy)Age<=21 Yrs (N=61) | Pre-B ALL Relapse <18 Mths From Dx (Chemotherapy) Age <=21 Yrs (N=49) | T-cell ALL (Chemotherapy) (N=22) | T-cell Lymphoblastic Lymphoma (LL) (Chemotherapy) (N=10)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 3 (3) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Anal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic necrosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 1 (1)
Peritoneal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Death NOS (General disorders) | 2 (2) | 24 (24) | 24 (24) | 9 (9) | 5 (5)
Fever (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Encephalitis infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 5 (5) | 3 (3) | 2 (2) | 1 (1)
Infective myositis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 8 (10) | 8 (8) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Cholesterol high (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 8 (8) | 1 (1) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 4 (4) | 1 (1) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 4 (4) | 2 (2) | 0 (0)
Akathisia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 8 (8) | 3 (3) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 4 (4) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 8 (8) | 5 (5) | 3 (3) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-B ALL Relapse < 36 Mths From Dx (Chemotherapy) Age >21 Yrs (N=4) | Pre-B ALL Relapse 18-36 Mths From Dx (Chemotherapy)Age<=21 Yrs (N=61) | Pre-B ALL Relapse <18 Mths From Dx (Chemotherapy) Age <=21 Yrs (N=49) | T-cell ALL (Chemotherapy) (N=22) | T-cell Lymphoblastic Lymphoma (LL) (Chemotherapy) (N=10)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 41 (47) | 27 (29) | 17 (17) | 7 (7)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 23 (23) | 22 (22) | 10 (10) | 2 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 7 (7) | 4 (4) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Rectal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 8 (8) | 3 (3) | 1 (1) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 11 (12) | 8 (8) | 4 (4) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 20 (22) | 15 (16) | 7 (8) | 4 (5)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 6 (6) | 1 (1) | 1 (1) | 2 (2)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periorbital infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Peritoneal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 6 (6) | 5 (5) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Splenic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 5 (5) | 2 (2) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 15 (15) | 8 (8) | 3 (3) | 3 (4)
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 8 (8) | 4 (4) | 3 (3) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibrinogen decreased (Investigations) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Forced expiratory volume decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GGT increased (Investigations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 7 (7) | 3 (3) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (3) | 16 (19) | 16 (21) | 5 (6) | 2 (2)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (3) | 39 (45) | 30 (34) | 18 (20) | 9 (10)
Platelet count decreased (Investigations) | 3 (4) | 44 (50) | 32 (39) | 18 (20) | 9 (10)
Serum amylase increased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 3 (3) | 38 (44) | 29 (31) | 12 (15) | 7 (9)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 6 (6) | 3 (3) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 10 (11) | 5 (5) | 3 (3) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 6 (6) | 3 (3) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 7 (9) | 5 (5) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 15 (16) | 13 (14) | 6 (6) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 6 (6) | 4 (4) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 7 (7) | 5 (5) | 0 (0) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 4 (4) | 6 (6) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less